CLINICAL TRIAL: NCT05650359
Title: A Randomized and Controlled Study of the Use of Orthopulse Photobiomodulation for Acceleration of Orthodontic Tooth Movement With Fixed Appliances
Brief Title: Study of the Use of Orthopulse Photobiomodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biolux Technology GmbH (Industry)
Collaborators: medXteam GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP_2021-02
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Orthodontics

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, open-label, multicenter PMCF study.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- OrthoPulse (Experimental): The study population includes a total of 41 patients (based on our sample size calculation), with 21 patients in group 1 and 21 patients in group 2. Eligible study participants are men and women over the age of 18 with permanent dentition who require orthodontic treatment.
  Interventions: Device: OrthoPulse
- Control (Active Comparator): The study population includes a total of 41 patients (based on our sample size calculation), with 21 patients in group 1 and 21 patients in group 2. Eligible study participants are men and women over the age of 18 with permanent dentition who require orthodontic treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: OrthoPulse — The OrthoPulse device is intended to accelerate orthodontic movement of teeth and reduce the overall treatment time for the patient. The device is intended to be used in conjunction with traditional orthodontic treatment with brackets and wires or aligners.
  OrthoPulse is an intra-oral (iO), Light Emitting Diode (LED) based, phototherapy device for the stimulation of metabolic activity of the alveolar bone, and the acceleration of orthodontic tooth movement during orthodontic treatment. The device uses safe, high-power LED arrays to produce photons at therapeutic wavelengths in the near infrared (nIR) portion of the light spectrum.
  OrthoPulse is an established device that uses low levels of light energy to stimulate the bone surrounding the roots of teeth and facilitate tooth movement which may reduce treatment time for braces or clear aligners.
  Arms: OrthoPulse
Other: No intervention — No intervention
  Arms: Control

SUMMARY:
This PMCF study evaluates the safety and performance of OrthoPulse photobiomodulation to accelerate tooth movement during alignment with fixed appliances.

DETAILED DESCRIPTION:
The purpose of the current clinical investigation performed in form of a post-market clinical follow-up (PMCF) study is to evaluate the performance of OrthoPulse by means of confirming the hypothesis that Subjects in the interventional group (group 1) will have a statistically significant average faster rate of tooth movement during the alignment phase than the average of subjects in the control group (group 2) (estimated 1.8x faster tooth movement) and to substantiate the clinical data for the application of OrthoPulse in case of fixed appliances (brackets).

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 18 years
* Indication for an orthodontic treatment with fixed appliances
* Presence of a written declaration
* Permanent dentition
* Class I-III malocclusion
* Between 4-10mm of crowding (estimated traditionally) in anterior teeth in mandibular arch (This will depend on the time we choose for the endpoint)

Exclusion Criteria:

* Simultaneous participation in another clinical investigation or study
* Prior participation in this study
* Persons who have been placed in an institution as a result of an administrative or judicial order
* Persons who are dependent on the sponsor, Investigator or the investigation site
* Anterior cross bite
* Spaces between anterior teeth
* Extractions or missing permanent teeth (except for third molars)
* No anticipated requirement of auxiliary appliances and/or elastics during treatment during alignment phase
* Acute oral infection or periodontal disease
* Active caries
* Pregnant patients or patients planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this PMCF study is the rate of tooth alignment. | 42 days after start of treatment
  The primary endpoint of this PMCF study is the rate of tooth alignment as per Little's irregularity index LII (measured as the distance of linear displacement in mm divided by a unit of time between the lower arch anterior 6 teeth) during the time between baseline and 42 days after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Dickerson, Principal Investigator — Private Practice 1200 W Warner Rd, Chandler, AZ 85224
Locations (1):
- Private Practice, Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: No